CLINICAL TRIAL: NCT02417012
Title: Does Intensive Life Style Intervention Reduce the Need for Glucose Lowering Medications in Patients With Type 2 Diabetes? The U-TURN Project
Brief Title: Lifestyle and Glucose Lowering Medication in T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TRYG Foundation (Other)
Responsible Party: Principal Investigator, Mathias Ried-Larsen, Group leader, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U-TURN
Record Dates: First submitted 2015-04-06; First posted 2015-04-15 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: lifestyle; exercise; physical activity; diet; glycemic control; hba1c; glucose lowering drugs
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- U-TURN intervention (Experimental): The intervention group will receive an intensive lifestyle intervention including partly supervised aerobic and strength exercise, diet plans and counseling by clinical dietitians. All exercise will be supervised initially and the supervision will be reduced gradually across the 12-month intervention. Additionally, the participants will be offered educational classes on implementation of a healthy lifestyle and diabetes education and support by trained nurses.
  Participants in this group will have their pharmacological treatment regulated by the study endocrinologists using a standardized pharmacological treatment. The treatment is in accordance with the Danish guidelines.
  Interventions: Behavioral: U-TURN
- Standard care (Active Comparator): The reference group will receive diabetes education and support by trained nurses.
  Participants in this group will have their pharmacological treatment regulated by the study endocrinologists using a standardized pharmacological treatment. The treatment is in accordance with the Danish guidelines.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: U-TURN — Participants in this group will receive individual and group based interventions on obtaining and maintaining a healthy lifestyle, while having the pharmacological treatment regulated
  Arms: U-TURN intervention
Behavioral: Standard care — Standard individual diabetes support
  Arms: Standard care

SUMMARY:
This study evaluates the effect of a lifestyle intervention maintenance of glycemic control while reducing glucose lowering drugs in patients with type 2 diabetes mellitus. The intervention group receives an intensive lifestyle intervention including exercise and diet lifestyle modifications. The reference group receives diabetes educational advice. Both groups will have their pharmacological treatment regulated across the study. The primary hypothesis is that lifestyle change is sufficient to maintain glycemic control while decreasing the anti-diabetic medication in a sample patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Adherence to lifestyle modifications including increased exercise and healthy diet improves glycemic control in patients with type 2 diabetes mellitus. However, few have investigated the combined effects of these lifestyle changes on maintenance of glycemic control while decreasing the usage of anti-diabetic medications.

The primary hypothesis is that lifestyle change is equivalent in maintaining glycemic control (Hba1c) compared to the standard pharmacological treatment,

The U-TURN trial also tests the effects on one key secondary outcome (glucose lowering medication) and examines the effects on sleep quality, fatigue sleepiness, sleep pattern, cardio vascular disease risk factors, psychological outcomes, blood pressure and cholesterol lowering medication. The participants (N=120) is randomized into a experimental group (N=80) and a standard care group (N=40).

Additionally, the effects of the study will be evaluated 24 month post randomization.

ELIGIBILITY:
Inclusion Criteria:

* Less than three anti-diabetic medications.
* Diabetes 2 duration of max 10 years
* BMI >25 but <40 kg/m2,
* Accept of medical regulation by the UTURN endocrinologists only
* Accept of purchasing a fitness club membership through U-TURN collaborator

Exclusion Criteria:

* Hba1c> 9% (75 mmol/mol)
* Insulin usage
* Presence of one or more of the following micro- and macrovascular complications of T2DM; a.Diabetic retinopathy (except mild nonproliferative retinopathy or early proliferative retinopathy) b. Macro-albuminuria or nephropathy c. Diabetic neuropathy (except mild affected vibratory testing (<50 Volt)) d. Arterial insufficiency e. Ischemic heart disease
* Steroid treatment (inhalation) until three months before the medical examination
* TSH raised/below the normal range
* Liver disease (ALAT/ASAT thrice normal range)
* Inability or contraindication to increased levels of physical activity (Pedersen BK and Saltin B)
* Evidence of anaemia
* Lung disease (except mild asthma and mild chronic obstructive pulmonary disease)
* Heart disease
* Kidney disease (creatinine above 130 µM or macro albuminuria)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Hba1c | 0, 3, 6, 9, 12 months
  blood sampling of Hba1c

SECONDARY OUTCOMES:
Change in glucose lowering medication | 0, 3, 6, 9, 12 months
  Change in doses of Metformin, GLP-1 analog, insulin. The change will be evaluate according to changes on the pre-specified regulation algorithm.

OTHER OUTCOMES:
incidence of hypo-glycemic episodes | 0, 3, 6, 9, 12, 24 months
  Self-report to study nurse
Changes Ldl cholesterol | 0, 3, 6, 9, 12, 24 months
  Blod sampling
Changes Hdl cholesterol | 0, 3, 6, 9, 12, 24 months
  Blood sampling
Changes total cholesterol | 0, 3, 6, 9, 12, 24 months
  Blood sampling
Changes in triglycerides | 0, 3, 6, 9, 12, 24 months
  Blood sampling
Changes in bdnf-a | 0, 12 months
  Blood sampling
Change in physical fitness | 0, 12, 24 months
  Progressive treadmill protocol
Change in body composition (DXA scan) | 0, 3, 6, 9, 12, 24 months
  DXA scan
Change in sleep quality | 0, 12, months
  Self-report using the PSQI questionnaire
Change in sleepiness | 0, 12, months
  Self-report using the Epsworth questionnaire
Change in sleep pattern | 0, 12, months
  Cardio-respiratory monitoring
Change in the degree of depression | 0, 12, 24 months
  Self-report using the BDI-II questionnaire
Change in Glucose tolerance (2-h oral glucose tolerance test) | 0, 12, 24 months
  2-h oral glucose tolerance test
Change in Well-being | 0, 12, 24 months
  Self-report using the questionnaire SF-36 and MFI20
Change in motivation for exercise | 0, 12, 24 months
  Self-report using the questionnaire BREQ-2
Change in cognitive function | 0, 12 months
  Self-report using the CANTAB test battery
Change in arterial function | 0, 12 months
  Arterial function will be determined using flow mediated dilation in a sub set of N=20 patients in each intervention arm (Total N=20)
Partial T2D remission | 24 months
  No active glucose lowering medication and HbA1c<48 mmol/mol and Fasting blood glucose<6,9 mmol/l
Full T2D remission | 24 months
  No active glucose lowering medication and HbA1c<39 mmol/mol and Fasting blood glucose<5.6 mmol/l
Change in low grade inflammation | 0, 12, 24 months
  The change in pro- and anti inflammatory markers will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ried-Larsen, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Center for Physical Activity Research, Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Pedersen BK, Saltin B. Evidence for prescribing exercise as therapy in chronic disease. Scand J Med Sci Sports. 2006 Feb;16 Suppl 1:3-63. doi: 10.1111/j.1600-0838.2006.00520.x. PMID 16451303
- [Derived] Legaard GE, Feineis CS, Johansen MY, Hansen KB, Vaag AA, Larsen EL, Poulsen HE, Almdal TP, Karstoft K, Pedersen BK, Ried-Larsen M. Effects of an exercise-based lifestyle intervention on systemic markers of oxidative stress and advanced glycation endproducts in persons with type 2 diabetes: Secondary analysis of a randomised clinical trial. Free Radic Biol Med. 2022 Aug 1;188:328-336. doi: 10.1016/j.freeradbiomed.2022.06.013. Epub 2022 Jun 25. PMID 35764194
- [Derived] Abildgaard J, Johansen MY, Skov-Jeppesen K, Andersen LB, Karstoft K, Hansen KB, Hartmann B, Holst JJ, Pedersen BK, Ried-Larsen M. Effects of a Lifestyle Intervention on Bone Turnover in Persons with Type 2 Diabetes: A Post Hoc Analysis of the U-TURN Trial. Med Sci Sports Exerc. 2022 Jan 1;54(1):38-46. doi: 10.1249/MSS.0000000000002776. PMID 34431828
- [Derived] MacDonald CS, Nielsen SM, Bjorner J, Johansen MY, Christensen R, Vaag A, Lieberman DE, Pedersen BK, Langberg H, Ried-Larsen M, Midtgaard J. One-year intensive lifestyle intervention and improvements in health-related quality of life and mental health in persons with type 2 diabetes: a secondary analysis of the U-TURN randomized controlled trial. BMJ Open Diabetes Res Care. 2021 Jan;9(1):e001840. doi: 10.1136/bmjdrc-2020-001840. PMID 33441418
- [Derived] Johansen MY, Karstoft K, MacDonald CS, Hansen KB, Ellingsgaard H, Hartmann B, Wewer Albrechtsen NJ, Vaag AA, Holst JJ, Pedersen BK, Ried-Larsen M. Effects of an intensive lifestyle intervention on the underlying mechanisms of improved glycaemic control in individuals with type 2 diabetes: a secondary analysis of a randomised clinical trial. Diabetologia. 2020 Nov;63(11):2410-2422. doi: 10.1007/s00125-020-05249-7. Epub 2020 Aug 20. PMID 32816096
- [Derived] MacDonald CS, Johansen MY, Nielsen SM, Christensen R, Hansen KB, Langberg H, Vaag AA, Karstoft K, Lieberman DE, Pedersen BK, Ried-Larsen M. Dose-Response Effects of Exercise on Glucose-Lowering Medications for Type 2 Diabetes: A Secondary Analysis of a Randomized Clinical Trial. Mayo Clin Proc. 2020 Mar;95(3):488-503. doi: 10.1016/j.mayocp.2019.09.005. Epub 2020 Jan 30. PMID 32007295
- [Derived] Johansen MY, MacDonald CS, Hansen KB, Karstoft K, Christensen R, Pedersen M, Hansen LS, Zacho M, Wedell-Neergaard AS, Nielsen ST, Iepsen UW, Langberg H, Vaag AA, Pedersen BK, Ried-Larsen M. Effect of an Intensive Lifestyle Intervention on Glycemic Control in Patients With Type 2 Diabetes: A Randomized Clinical Trial. JAMA. 2017 Aug 15;318(7):637-646. doi: 10.1001/jama.2017.10169. PMID 28810024
- [Derived] Ried-Larsen M, Christensen R, Hansen KB, Johansen MY, Pedersen M, Zacho M, Hansen LS, Kofoed K, Thomsen K, Jensen MS, Nielsen RO, MacDonald C, Langberg H, Vaag AA, Pedersen BK, Karstoft K. Head-to-head comparison of intensive lifestyle intervention (U-TURN) versus conventional multifactorial care in patients with type 2 diabetes: protocol and rationale for an assessor-blinded, parallel group and randomised trial. BMJ Open. 2015 Dec 9;5(12):e009764. doi: 10.1136/bmjopen-2015-009764. PMID 26656025